CLINICAL TRIAL: NCT00864526
Title: A Relative Bioavailability Study of Oxycodone 5 mg / Ibuprofen 400 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B0605001
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Oxycodone; Ibuprofen; Healthy subjects
MeSH Terms: interventions — Oxycodone; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Oxycodone HCl 5 mg / Ibuprofen 400 mg tablets, single dose
  Interventions: Drug: Oxycodone HCl 5 mg / Ibuprofen 400 mg tablets, single dose
- B (Active Comparator): COMBONOX® tablets, single dose
  Interventions: Drug: COMBONOX® tablets, single dose

INTERVENTIONS:
Drug: Oxycodone HCl 5 mg / Ibuprofen 400 mg tablets, single dose — A: Experimental SSubjects received Actavis formulated products under fasting conditions
  Other Names: Oxycodone; Ibuprofen
  Arms: A
Drug: COMBONOX® tablets, single dose — B: Active comparator Subjects received Forest Pharmaceuticals, Inc formulated products under fasting conditions
  Other Names: Oxycodone; Ibuprofen
  Arms: B

SUMMARY:
To compare the relative bioavailability of oxycodone HCl 5 mg / ibuprofen 400 mg tablets (Actavis Elizabeth LLC, Lot No. PI-1565) with that of COMBONOX® tablets (Forest Pharmaceuticals, Inc., Lot No. 010550) in healthy adult volunteers under fasting conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Single dose randomized, two-period, two-treatment, two-sequence crossover study under fasting conditions comparing equal doses of the test and reference products.

Official Title: A Relative Bioavailability Study of Oxycodone 5 mg / Ibuprofen 400 mg Tablets Under Fasting Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. All subjects selected for this study will be at least 18 years of age.
2. Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.

Each female subject will be given a serum pregnancy test as part of the pre-study screening process.

At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.

Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.

Clinical laboratory measurements will include the following as a minimum:

Hematology: hemoglobin, hematocrit, red blood cell count, platelets, and white blood cell count (with differential).

Clinical Chemistry: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase.

Urine Analysis: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells.

HIV Screen: (pre-study only)

Hepatitis-B, C Screen: (pre-study only)

Drugs of Abuse Screen: (pre-study and at check-in each dosing period)

Electrocardiograms of all participating subjects will be recorded before initiation of the study and filed with each subject's case report forms.

Exclusion Criteria:

1. Subjects with a history of alcoholism or drug addiction (during past 2 years), or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (during past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study. [Subjects who have had a cholecystectomy will not be eligible unless approved by the sponsor.]
2. Subjects whose clinical laboratory test values are outside the reference range may be retested at the discretion of the clinical investigator. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
3. Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study.
4. All subjects will have urine/saliva samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at check-in each dosing period. Subjects found to have urine/saliva concentrations of any of the tested drugs will not be allowed to participate.
5. Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
6. Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
7. Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives anytime during the 6 months prior to study dosing, or used oral hormonal contraceptives or a contraceptive transdermal patch within 14 days before dosing will not be allowed to participate.
8. All female subjects will be screened for pregnancy prior to dosing each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
9. Subjects with positive HIV or hepatitis screen will not be allowed to participate in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Longnecker,, M.D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research, Inc, Saint Charles, Missouri, United States